CLINICAL TRIAL: NCT00534157
Title: Intraocular Pressure as a Predictor of Intracranial Pressure in the Acutely Head-Injured Population
Brief Title: Study of Eye Pressure as a Predictor of Intracranial Pressure in the Acutely Head-Injured Population
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Other Study IDs: 2004H0126
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-03

CONDITIONS: Craniocerebral Trauma
Keywords: intracranial pressure; intraocular pressure; tonometry
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the pressure in the eye of a severely head-injured person correlates with the pressure in the person's skull. This is a prospective study of patients aged 18 and older who have experienced a traumatic closed head injury and are intubated either before or during the time they are in the Emergency Department (ED). Identified patients have an eye pressure measurement performed in the trauma bay by an OSU ED physician not involved in their care. Information about their hospital stay, including the first brain pressure measurement if a such a measuring device is used, will be collected. In addition, the outcome of their hospital stay will be recorded.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of morbidity and mortality in the United States, with an estimated 1.5 million American sustaining a TBI and 50,000 people dying from a TBI each year. While the immediate, or primary, injury causes significant damage, secondary injury is caused by cerebral edema, increased intracranial pressure, and resultant hypoperfusion and ischemia. Elevated intracranial pressure is strongly associated with poor recovery and death; failure to control intracranial pressure is likewise associated with poor outcomes and mortality.

Early detection of elevated ICP allows for the initiation of early therapy. However, patients with significant head injuries are often intubated for airway protection. The sedation required for intubation obscures the ED neurologic exam. Precise measurement of elevated ICP has required invasive monitoring via ventriculostomy. Yet this method is only provided at set institutions with neurosurgical services. Further there are distinct time delays between the trauma occurrence, transportation to a facility with neurosurgical services and placement of ventriculostomies. There is at the forefront, then, to establish non-invasive measures of ICP that are both time efficient and reliable.

Previous studies, including a pilot study conducted at this institution, showed a correlation between intraocular and intracranial pressure. However, this relationship has not been tested in an acute care trauma setting. We propose an observational cohort study of critically injured trauma patients with suspected closed head injury. Patients requiring intubation and mechanical ventilation pose a significant challenge to assess neurologically, as they are almost always sedated and often chemically paralyzed to facilitate airway management. Therefore, it is in this population of intubated trauma patients with suspected head injury that we will evaluate the use of tonometry to predict intracranial pressure from intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute traumatic head injury
* Intubated prior to arrival in the Emergency Department or in the Emergency Department, including patients transferred from other facilities

Exclusion Criteria:

* Too unstable to allow the investigator access to the head of the bed to perform tonometry.
* Severe ocular or facial trauma such that an intact globe is not accessible
* Known history of glaucoma
* Penetrating head injury
* Patients that undergo operative decompression prior to the placement of an intracranial pressure monitor may be screened in the trauma bay and have an intraocular pressure obtained; however, these patients will not be included in the intraocular / intracranial pressure analysis.
* Known allergy to latex or tetracaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-06; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Hiestand, MD, Principal Investigator — The Ohio State University Department of Emergency Medicine
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States